CLINICAL TRIAL: NCT03661424
Title: A Phase I Study of Anti-CD3 x Anti-Her2/Neu (Her2Bi) Armed Activated T Cells (ATC) in Patients With Breast Cancer Leptomeningeal Metastases
Brief Title: BATs in Patients With Breast Cancer and Leptomeningeal Metastases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow study accrual, partially due to pandemic
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Camilo E. Fadul, MD, Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20805
Record Dates: First submitted 2018-08-22; First posted 2018-09-07 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer Female; Leptomeningeal Metastases
Keywords: Metastatic Breast Cancer; Adoptive Cell Therapy; Armed Activated T-cells; Bispecific Antibodies; Immunotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Test dose then 8 doses HER2 Bi-armed activated T-cells (BATs) (Experimental): Approximately 4 weeks following registration and blood collection, participants are given a test dose of HER2 BATs followed by 8 weekly infusions. Infusions are given intraventricularly.
  Interventions: Drug: HER2 BATs

INTERVENTIONS:
Drug: HER2 BATs — A test dose (1 million cells) of HER2 BATs (at one of the two dose levels: 5 million cells or 10 million cells per infusion) followed by 8 weekly infusions of Her2 BATs delivered into the ventricle of the brain. Infusions are delivered weekly over 8 weeks with brain MRIs prior to first infusion and following the eighth infusion. Blood will be drawn for immune evaluation before during and after study treatment.

SUMMARY:
This study uses bi-specific antibody (HER2Bi) armed activated T-cells (HER2 BATs) to target breast cancer cells that have metastasized to the membranes surrounding the brain and spinal cord. This is known as leptomeningeal metastases. Two doses will be evaluated in order to determine a safe dose.

Study treatment includes a test dose of HER2 BATs followed by 8 weekly infusions of HER2 BATs at the assigned dose level. Before, during and after study treatment, participants will be monitored objectively by brain MRIs and clinically through physical and neurological exams, and blood and cerebrospinal fluid will be collected to evaluate immune responses.

DETAILED DESCRIPTION:
Once subjects are determined eligible, white blood cells (lymphocytes) are collected via leukapheresis procedure approximately 3 to 4 weeks prior to the first BATs infusion. The white blood cells, specifically T cells, are then mixed with two proteins in order to activate the cells to multiply.

After approximately 14 days in culture, the activated T cells are coated with OKT3 and trastuzumab/Herceptin (HER2Bi), and washed to remove excess Herceptin in order to produce bispecific antibody armed T cells (BATs). Cells are then frozen and stored until scheduled to be infused.

Up to 2 weeks following leukapheresis, participants will undergo surgery to place the catheter/reservoir into the lateral ventricle of the brain to allow intraventricular administration of HER2 BATs and a chemotherapy agent methotrexate. A few weeks later, participants will receive the intraventricular methotrexate in order to control disease while the BATs product is being manufactured. About 4-5 weeks following the leukapheresis and at least 7 days after receiving methotrexate, study treatment will begin with a test dose of HER2 BATs. If this dose is well tolerated by the participant, she will then receive 8 weekly doses of HER2 BATs at the assigned dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Participants must be female.
3. Histologically confirmed breast cancer (any Her2, estrogen receptor (ER), or progesterone receptor (PR) expression) with leptomeningeal metastasis (LM) as determined by imaging and/or cerebrospinal fluid (CSF) cytology.
4. 18 years of age or older.
5. Women of reproductive potential must agree to use an effective method of contraception during therapy. Effective methods include intrauterine device (IUD), vasectomy of the male partner, diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, or hormonal contraceptive.
6. Karnofsky Performance Status (KPS) of ≥60.
7. Eligible for intraventricular (IVENT) catheter/reservoir placement as determined by neurosurgery.
8. Demonstrate adequate organ function as defined below. All screening labs should be performed within 10 days of confirmation of eligibility.

Absolute lymphocyte count ≥ 500/mm3 Absolute neutrophil count ≥ 1000/mcL Platelets ≥ 100,000 / mnL Hemoglobin ≥ 8 g/dL BUN ≤ 1.5 x upper limit of normal (ULN) Serum creatinine within the normal limits OR measured or calculated creatinine clearance ≥ 60 mL/min 1.73m2 Serum total bilirubin ≤ 2 x ULN OR AST (SGOT) and ALT (SGPT) ≤ 5 x ULN Albumin ≥ 2.5 mg/dL

Exclusion Criteria:

1. Current severe increased intracranial pressure with clinical or imaging findings suggestive of herniation, status epilepticus, or other serious complications requiring emergency or urgent intervention.
2. Patients who cannot have MRI studies for any reason (intolerance, medical contraindication, etc.).
3. Patients with a history of another malignancy within 1 year of study enrollment with the following exceptions: patients with history of ductal carcinoma in situ (DCIS), squamous cell skin cancers, or other in situ carcinomas are not excluded.
4. Patients with unresolved autoimmune toxicity.
5. Patients with a known disorder that increases the risk of bleeding (e.g., Hemophilia, von Willebrands disease, or clinically significant clotting factor deficiency).
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Administration of any investigational agents, immunomodulating agents, radiation therapy or chemotherapy for MBC within the 7 days before the 80 mL blood draw to collect cells for study treatment.
8. Has Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
9. Pregnancy or lactation at the time of registration.
10. Psychiatric or addictive disorders or other conditions that in the opinion of the investigator would preclude the patient from complying with the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Types of adverse events (AEs) | For each participant, AEs will be collected from the time of the first protocol-related procedure through 30 days following last infusion of BATs. SAEs considered related to study treatment will also be collected following this period.
  Types of any adverse events or abnormalities of laboratory tests
Frequency of adverse events (AEs) | For each participant, AEs will be collected from the time of the first protocol-related procedure through 30 days following last infusion of BATs. SAEs considered related to study treatment will also be collected following this period.
  Frequency of any adverse events or abnormalities of laboratory tests
Severity of adverse events (AEs) | For each participant, AEs will be collected from the time of the first protocol-related procedure through 30 days following last infusion of BATs. SAEs considered related to study treatment will also be collected following this period.
  Severity of any adverse events or abnormalities of laboratory tests
Timing of onset of adverse events | For each participant, AEs will be collected from the time of the first protocol-related procedure through 30 days following last infusion of BATs. SAEs considered related to study treatment will also be collected following this period.
  Timing of onset of any adverse events or abnormalities of laboratory tests
Duration of adverse events | For each participant, AEs will be collected from the time of the first protocol-related procedure through 30 days following last infusion of BATs. SAEs considered related to study treatment will also be collected following this period.
  Duration of any adverse events or abnormalities of laboratory tests
Relationship to study therapy of any adverse events or abnormalities of laboratory tests as determined by CTCAE v5.0 will be assessed based on protocol-defined relationships of definitely, probably, possibly, unlikely and unrelated to study therapy. | For each participant, AEs will be collected from the time of the first protocol-related procedure through 30 days following last infusion of BATs. SAEs considered related to study treatment will also be collected following this period.
  Relationship to study therapy of any adverse events or abnormalities of laboratory tests
Number of participants achieving at least 80% of the planned HER2 BATs dose. | An average of 4 weeks following blood draw to collect cells for HER2 BATs
  If at least 80% of the planned dose of cells cannot be produced for 3 consecutive participants at a designated dose level, that dose level will be considered not feasible.

SECONDARY OUTCOMES:
Immune shift: in vitro cytotoxicity assays and/or IFN-y EliSpots against breast cancer cell lines | Blood for immune analysis collected prior to, during and following study treatment (tx) (up to 6 months following study tx).
  Immune shift induced by Her2 BATs as detected by in vitro cytotoxicity assays and/or IFN-γ EliSpots against breast cancer cell lines
Immune shift: Phenotyping of activating and regulatory immune cells | Blood for immune analysis collected prior to, during and following study treatment (tx) (up to 6 months following study tx).
  Immune shift induced by Her2 BATs as detected by phenotyping of activating and regulatory immune cells
Immune shift: Measurement of cytokine patterns | Blood for immune analysis collected prior to, during and following study treatment (tx) (up to 6 months following study tx).
  Immune shift induced by Her2 BATs as detected by measurement of cytokine patterns
Immune shift: Determination of anti-Her2 antibodies | Blood for immune analysis collected prior to, during and following study treatment (tx) (up to 6 months following study tx).
  Immune shift induced by Her2 BATs as detected by determination of anti-Her2 antibodies
Correlation of clinical and immune response characteristics to progression-free survival | Blood collected prior to, during and following study treatment (tx) (up to 6 months following study tx). Clinical characteristics and imaging prior to and after study tx through 1st progression
  Correlation individually and by heatmap analysis of imaging, pathology, clinical, and immune response characteristics to progression free survival (PFS)
Correlation of clinical and immune response characteristics to overall survival | Blood for immune analysis collected prior to, during and after study treatment (tx) (up to 6 months following study tx). Clinical characteristics and imaging prior to and after study tx through 1st progression
  Correlation individually and by heatmap analysis of imaging, pathology, clinical, and immune response characteristics to overall survival (OS).
Objective response rate (ORR) | Assessed on MRI studies done 9 weeks after first BATs infusion
  Proportion of participants with complete or partial response according to brain and spine MRI
Progression-free survival (PFS) | From date of first BATs infusion (approximately 4 weeks following eligibility confirmation) until the date of confirmed progression, assessed up to 28 months
  Length of time from study participation initiation through disease progression for each participant
Overall survival (OS) | Through each participant's death or for 2 years following study treatment
  Length of time from study participation initiation through death or for 2 years following study treatment for each participant
MD Anderson Symptom Inventory for Spinal Tumors (MDASI - SP) | Prior to test dose of study treatment, prior to the 5th and 8th weekly infusions, and 30 days following last infusion
  The MDASI- SP is a 24 item questionnaire that focuses on symptoms related to spinal tumors. For each potential symptom, there is an eleven-point scale where 0 is "Not Present" and 10 is "As Bad As You Can Imagine" so the minimum score would be 0 and the maximum score would be 240. For a subset of questions, the scale measures how much the symptoms interfered with other parts of life and the scale ranges from symptoms that "Did Not Interfere" (0) to those that "Interfered Completely" (10). Lower scores indicate fewer/less severe/less interfering symptoms and higher scores indicate more/more severe/more interfering symptoms.
MD Anderson Symptom Inventory for Brain Tumors (MDASI- BT) | Prior to test dose of study treatment, prior to the 5th and 8th weekly infusions, and 30 days following last infusion
  The MDASI- BT is a 28 item questionnaire that focuses on symptoms related to brain tumors. For each potential symptom, there is an eleven-point scale where 0 is "Not Present" and 10 is "As Bad As You Can Imagine" so the minimum score would be 0 and the maximum score would be 280. For a subset of questions, the scale measures how much the symptoms interfered with other parts of life and the scale ranges from symptoms that "Did Not Interfere" (0) to those that "Interfered Completely" (10). Lower scores indicate fewer/less severe/less interfering symptoms and higher scores indicate more/more severe/more interfering symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Fadul, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum LG, Thakur A, Al-Kadhimi Z, Colvin GA, Cummings FJ, Legare RD, Dizon DS, Kouttab N, Maizel A, Colaiace W, Liu Q, Rathore R. Targeted T-cell Therapy in Stage IV Breast Cancer: A Phase I Clinical Trial. Clin Cancer Res. 2015 May 15;21(10):2305-14. doi: 10.1158/1078-0432.CCR-14-2280. Epub 2015 Feb 16. PMID 25688159
- [Background] Vaishampayan U, Thakur A, Rathore R, Kouttab N, Lum LG. Phase I Study of Anti-CD3 x Anti-Her2 Bispecific Antibody in Metastatic Castrate Resistant Prostate Cancer Patients. Prostate Cancer. 2015;2015:285193. doi: 10.1155/2015/285193. Epub 2015 Feb 23. PMID 25802762